CLINICAL TRIAL: NCT07097935
Title: A Phase Ib/II Clinical Study Evaluating the Safety, Efficacy, Tolerability, and Pharmacokinetics of HS-10516 Combination Therapy in Patients With Advanced Renal Cell Carcinoma
Brief Title: Study of HS-10516 Combination Therapy in Patients With Advanced Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10516-103
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ib (Dose exploration phase) Phase II (Proof-of-concept phase) (Experimental): Treatment cycles are set at 28 days, with investigational product administration continuing until disease progression or meeting other treatment discontinuation criteria.
  Interventions: Drug: HS-10516 + Lenvatinib

INTERVENTIONS:
Drug: HS-10516 + Lenvatinib — Administered orally.

SUMMARY:
This is a multicenter, open-label, Phase Ib/II clinical study evaluating the safety, efficacy, tolerability, and pharmacokinetic/pharmacodynamic (PK/PD) profiles of HS-10516 in combination with lenvatinib in patients with advanced clear cell renal cell carcinoma (ccRCC) who have progressed after receiving at least one prior line of systemic therapy. The study comprises two distinct phases: a dose exploration phase and a proof-of-concept phase.

DETAILED DESCRIPTION:
The study will commence with a dose exploration phase employing a safety lead-in approach. Treatment cycles are set at 28 days, with investigational product administration continuing until disease progression or meeting other treatment discontinuation criteria. Each dose level will enroll 3-6 participants for dose-limiting toxicity (DLT) assessment to evaluate the tolerability, safety, and PK/PD profiles of HS-10516 combined with lenvatinib. The Safety Review Committee (SRC) will determine subsequent dose levels for exploration through joint deliberation. If all predefined dose levels prove intolerable, the SRC may authorize exploration of lower dose levels. Additionally, PK expansion cohorts (up to 12 participants per cohort) may be implemented in suitable dose levels.

Following identification of safe dose levels in the exploration phase, 1-2 dose cohorts will advance to the proof-of-concept phase, with each cohort enrolling up to 40 participants to further assess therapeutic efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Histologically confirmed unresectable, locally advanced or metastatic clear cell renal cell carcinoma (ccRCC) with disease progression during or after receiving ≥1 prior line of systemic therapy in the advanced setting.
3. Patients have at least one target lesion according to RECEST 1.1. The requirements for target lesions are: measurable lesions without local treatment such as irradiation, or with definite progress after local treatment, with the longest diameter ≥ 10 mm in the baseline period (in case of lymph nodes, the shortest axis ≥ 15 mm is required). Patients with only brain and/or bone lesions as target lesions will not be included.
4. ECOG performance status was 0-1 and did not deteriorate in the previous 2 weeks.
5. Estimated life expectancy greater than (>) 12 weeks.
6. Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 12 months after the last dose. Likewise, men also consent to use adequate contraceptive method within the same time limit.
7. Females must have the evidence of non-childbearing potential
8. Sign informed consent form.

Exclusion Criteria:

1. Prior or Current Treatments:

   1. Previous or current use of hypoxia-inducible factor inhibitors.
   2. Previous or current use of lenvatinib.
   3. Use of Chinese herbal medicine with antitumor indications within 2 weeks prior to the first dose or requirement for such treatment during the study.
   4. Administration of cytotoxic chemotherapy or other systemic antitumor therapies (e.g., endocrine therapy, molecular targeted therapy) within 2 weeks or 5 half-lives (whichever is shorter) prior to the first dose, or requirement for such treatments during the study.
   5. Use of large-molecule antitumor drugs within 4 weeks prior to the first dose or requirement for such treatment during the study.
   6. Use of CYP2C19 strong inhibitors/inducers or narrow therapeutic index sensitive substrates within 7 days prior to the first dose, or requirement for continued use during the study.
   7. Local radiotherapy (except brain radiotherapy; see Criterion 6) within 2 weeks prior to the first dose, or >30% bone marrow irradiation/large-field radiotherapy within 4 weeks prior to the first dose.
   8. Major surgery (e.g., craniotomy, thoracotomy, laparotomy; Grade 3/4 per Chinese Medical Technical Clinical Application Regulations) within 4 weeks prior to the first dose.
   9. Participation in other interventional clinical trials within 4 weeks prior to the first dose or within 5 half-lives of investigational drugs (whichever is longer).
2. Resting pulse oximetry <92% at screening.
3. Severe pulmonary dysfunction requiring intermittent/long-term oxygen therapy.
4. Unresolved Grade >1 toxicities from prior anti-tumor therapy (per CTCAE v5.0).
5. History of second primary malignancy.
6. Known or suspected active CNS metastases/leptomeningeal disease.
7. Inadequate bone marrow reserve or serious organ dysfunction.
8. Severe, uncontrolled, or active cardiovascular disease.
9. Severe or poorly controlled diabetes.
10. Severe or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: MTD or RP2D | Up to 3 months
  MTD or RP2D was determined by number of participants with DLT in dose levels. A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0).
Phase II: Objective Response Rate (ORR) | Up to 12 months.
  The percentage of patients who have achieved complete response and partial response, according to response evaluation criteria in solid tumors (RECIST) 1.1 by investigator's assessment.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Up to 36 months.
  Incidence of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Disease control rate (DCR) | Up to 24 months.
  The percentage of patients who have achieved complete response, partial response, and stable disease, according to response evaluation criteria in solid tumors (RECIST) 1.1 by investigator's assessment.
Duration of response (DoR) | Up to 24 months.
  The time from complete or partial response to disease progression or death, according to response evaluation criteria in solid tumors (RECIST) 1.1 by investigator's assessment.
Progression-free survival (PFS) | Up to 24 months.
  Progression free survival is defined as the duration of time from study entry to time of progression, death, or is censored at date of last disease assessment.
Overall survival (OS) | Up to 3 years.
  Overall survival is defined as the duration of time from study entry to death or the date of last contact.
Maximum plasma concentration (Cmax) | Up to 24 months.
  Cmax is defined as maximum observed serum concentration obtained directly from the observed concentration-time data.
Time of maximum concentration (Tmax) | Up to 24 months.
  Tmax is defined as the time required for a drug to reach peak concentration in plasma.
AUC0-t | Up to 24 months.
  Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China